CLINICAL TRIAL: NCT06622187
Title: Bleeding Prevention With Desmopressin for Allograft Kidney Biopsies: a Double-blind Randomized Study
Brief Title: Bleeding Prevention With Desmopressin for Allograft Kidney Biopsies
Acronym: BRIDGE
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0270
Record Dates: First submitted 2024-09-03; First posted 2024-10-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Bleeding; Transplant, Kidney; Desmopressin; Kidney Biopsy
MeSH Terms: conditions — Hemorrhage | interventions — Deamino Arginine Vasopressin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Chloride (Placebo Comparator)
  Interventions: Drug: Sodium Chloride
- Desmopressin (DDAVP) (Experimental)
  Interventions: Drug: Desmopressin (DDAVP)

INTERVENTIONS:
Drug: Desmopressin (DDAVP) — Patients in the intervention group will receive desmopressin 0.3ug/kg administered as an intravenous infusion 1h before the proposed procedure
  Arms: Desmopressin (DDAVP)
Drug: Sodium Chloride — Patients in the control group will receive sodium chloride 0.9% 100mL administered as an intravenous infusion 1h before the proposed procedure
  Arms: Sodium Chloride

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of desmopressin to prevent bleeding after percutaneous renal graft biopsy in patients at high risk of bleeding.

Researchers will compare desmopressin (DDAVP) to placebo to see if the drug reduces the risk of bleeding events related to kidney biopsy.

Participants will receive intravenous desmopressin medication (100ml) or placebo (100mL of saline solution) before the kidney biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients with GFR <60ml/min/1,73m²
* Need for graft biopsy as indicated by the kidney transplant medical team
* Platelets >80.000 cells/mm³
* Blood pressure levels controlled before the procedure
* Normal coagulogram levels

Exclusion Criteria:

* Pregnant women
* Prior history of allergic reaction to DDAVP
* Use of prohibitive medications in screening: warfarin, direct oral anticoagulants, unfractionated and low molecular weight heparin in full anticoagulation doses
* History of previous blood dyscrasias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Bleeding events | Immediately post-biopsy until 48 hours post-biopsy
  Incidence of bleeding related to the procedure

SECONDARY OUTCOMES:
Major bleeding | Immediately post-biopsy until 48 hours post-biopsy
  Incidence of major bleeding, defined as need for transfusion of blood components, need for embolization, nephrectomy or procedure-related death
Minor bleeding | Immediately post-biopsy until 48 hours post-biopsy
  Incidence of minor bleeding, defined as presence of macroscopic hematuria, hematoma on ultrasound 24 hours post-procedure or drop in hemoglobin greater than 20%

OTHER OUTCOMES:
Number of participants with hyponatremia, skin reaction, anaphylaxis | Immediately pre-biopsy until 24 hours post-biopsy
  Number of participants with hyponatremia, skin reaction, anaphylaxis [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bauer, MD, PhD, Principal Investigator — Hospital Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
it is not known whether there will be a plan to make IPD available.

REFERENCES:
- [Background] Sethi J, Bansal S, Lal A, Kohli HS, Rathi M. Role of Desmopressin Acetate before Percutaneous Ultrasound-Guided Kidney Biopsy in Patients with Kidney Dysfunction. Indian J Nephrol. 2024 May-Jun;34(3):228-232. doi: 10.4103/ijn.ijn_34_23. Epub 2023 Sep 29. PMID 39114394
- [Background] Leclerc S, Nadeau-Fredette AC, Elftouh N, Lafrance JP, Pichette V, Laurin LP. Use of Desmopressin Prior to Kidney Biopsy in Patients With High Bleeding Risk. Kidney Int Rep. 2020 May 20;5(8):1180-1187. doi: 10.1016/j.ekir.2020.05.006. eCollection 2020 Aug. PMID 32775817
- [Background] Sattari SA, Shahoori A, Shahbazian H, Sabetnia L, Aref A, Sattari AR, Ghorbani A. Desmopressin Acetate in Percutaneous Ultrasound-Guided Native Kidney Biopsy in Patients with Reduced Kidney Function: A Double-Blind Randomized Controlled Trial. Iran J Kidney Dis. 2022 Jul;16(4):238-245. PMID 35962638
- [Background] Manno C, Bonifati C, Torres DD, Campobasso N, Schena FP. Desmopressin acetate in percutaneous ultrasound-guided kidney biopsy: a randomized controlled trial. Am J Kidney Dis. 2011 Jun;57(6):850-5. doi: 10.1053/j.ajkd.2010.12.019. Epub 2011 Feb 26. PMID 21354681
- [Background] Mannucci PM, Remuzzi G, Pusineri F, Lombardi R, Valsecchi C, Mecca G, Zimmerman TS. Deamino-8-D-arginine vasopressin shortens the bleeding time in uremia. N Engl J Med. 1983 Jan 6;308(1):8-12. doi: 10.1056/NEJM198301063080102. PMID 6401193